CLINICAL TRIAL: NCT00585676
Title: Impact of Antenatal Betamethasone on Plasma Glucose Levels
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Deborah A. Wing, Professor and Director, Maternal-Fetal Medicine, University of California, Irvine
Other Study IDs: 436-07
Record Dates: First submitted 2008-01-02; First posted 2008-01-03 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Diabetic: Patients with Diabetes
- Abnormal glucose level: Patients who were screened and had abnormal blood glucose levels
- Control: Non-diabetic (normal glucose screening)

SUMMARY:
It is known that administration of steroids increases blood sugar levels. Administration of betamethasone is common practice during pregnancy to women at risk for preterm delivery. However, it is unknown the magnitude of the changes in glucose these women have after receiving betamethasone. The purpose of this study is to determine the magnitude and timing of the increase in blood sugar in pregnant women without diabetes who receive steroids.

DETAILED DESCRIPTION:
There is a substantial body of evidence that the administration of corticosteroids to patients deemed to be at risk for preterm delivery (delivery prior to 37 weeks gestation) decreases the risk of respiratory distress syndrome, intraventricular hemorrhage, and neonatal death. Current recommendations from the National Institute of Health (NIH) and the American College of Obstetricians and Gynecologists (ACOG) are that patients with pregnancies that are between 24-34 weeks gestation deemed at risk for preterm delivery receive antenatal corticosteroids. The recommended dosing is two doses of betamethasone 12 mg given 24 hours apart as an intramuscular injection. (Alternatively, dexamethasone 6 mg given intramuscularly every 6 hours for 4 doses may be administered. Betamethasone is used preferentially in our institution.)

Glucocortiocoids have a well-known effect on glucose metabolism. They increase blood glucose levels by antagonizing insulin and decreasing synthesis of insulin, thus inhibiting peripheral glucose utilization and increasing gluconeogenesis (the process by which the body produces glucose). Pregnancy is also characterized by a relative insulin resistance that results in glucose intolerance. It follows, then, that the combination of pregnancy and corticosteroids could cause significant disruption of glucose homeostasis.

Routinely in pregnancy, gestational diabetes is diagnosed by the administration of a glucose tolerance test consisting of ingestion of 50g of glucose followed by a serum glucose level one hour later. This is known as a one-hour post-glucola test. A value of 140 mg/dL is considered abnormal, and prompts administration of the 3-hour glucose tolerance test. This test consists of a fasting blood sugar, followed by serum glucose levels after a 100g oral glucose challenge at 1-, 2- and 3-hours. A profile with two or more abnormal values is considered diagnostic for gestational diabetes. In 1997 Fisher et al retrospectively compared the incidence of gestational diabetes in those patients who had received tocolytics and antenatal corticosteroids to those who did not, and found a higher incidence of both abnormal one-hour glucose screening tests and gestational diabetes in those patients who received steroids and tocolytics (medications used to try to decrease uterine contractions). However, the interval between the receipt of steroids and the administration of the glucose screening test was quite variable in this study. Shelton et al in 2002 evaluated the extent of hyperglycemia in non-diabetic patients who received multiple weekly doses of corticosteroids. They found that the fasting glucose levels increased for several days following the first course of steroids, returned to normal, and then remained persistently elevated in those patients who received three or more courses. Postprandial levels were not significantly altered. A study by Gurbuz et al in 2003 assessed the effects of betamethasone on the one-hour glucola test and found that although there was an initial effect on the screening test, this effect was transient and resolved generally one week after the administration of the second dose of betamethasone. These patients had a one-hour screening test performed prior to the administration of corticosteroids. The dosing regimen of betamethasone, however, was different from that recommended by ACOG. Thus far, no study has reported if: (1) there is significant hyperglycemia in non-diabetic patients who receive corticosteroids and (2) how the magnitude and pattern of the increase in glucose differs in patients with normal and abnormal one-hour glucolas or with diabetes. This study will be conducted as a pilot study, as there is no reports of the extent of hyperglycemia that occurs in non-diabetic patients after administration of corticosteroids to guide a sample size calculation. We will plan to obtain thirty non-diabetic subjects with fifteen diet-controlled diabetic controls for comparison. The hypothesis is that those patients that are not diabetic will not have the same extent of hyperglycemia as those who are diabetic.

ELIGIBILITY:
Inclusion criteria:

* Candidates for antenatal corticosteroids (including gestational age between 24-34 weeks)

Exclusion criteria:

* Age less than 18 years
* Pre-existing maternal corticosteroid or beta-mimetic tocolytic use
* Pre-gestational diabetes mellitus, class C or greater
* Pre-existing adrenal or pancreatic dysfunction
* Evidence of infection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women receiving corticosteroids
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve of blood glucose | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Nageotte, MD, Principal Investigator — Miller Children's Hospital
Locations (1):
- Miller Children's Hospital, Long Beach, California, United States